CLINICAL TRIAL: NCT05517928
Title: Exploratory Study of the Impact of Lactobacillus Rhamnosus GG on Proton Pump Inhibitor-Induced Gut Dysbiosis
Brief Title: A Study to Evaluate the Impact of Lactobacillus Rhamnosus GG on Proton Pump Inhibitor-Induced Gut Dysbiosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John K. DiBaise, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 21-007621
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Healthy
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus rhamnosus GG Group (Experimental): Subjects will receive omeprazole daily for 56 days. After 28 days, subjects will receive Lactobacillus rhamnosus GG two capsules daily taken with a meal.
  Interventions: Drug: Omeprazole; Dietary Supplement: Lactobacillus rhamnosus GG
- Placebo Group (Placebo Comparator): Subjects will receive omeprazole daily for 56 days. After 28 days, subjects will receive placebo two capsules daily taken with a meal.
  Interventions: Drug: Omeprazole; Drug: Placebo

INTERVENTIONS:
Drug: Omeprazole — 40 MG oral capsules daily
Dietary Supplement: Lactobacillus rhamnosus GG — Given as Culturelle Digestive Probiotic in the form of oral capsules daily
  Arms: Lactobacillus rhamnosus GG Group
Drug: Placebo — Oral capsules daily that look exactly like the study drug, but contains to active ingredient
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to investigate the impact of the probiotic Lactobacillus rhamnosus (LGG) on proton pump inhibitor (PPI)-induced changes to the microbes that live in the gastrointestinal tract and are passed out in the stool. PPI medicines reduce stomach acid and are commonly used to treat acid reflux disease.

ELIGIBILITY:
Inclusion Criteria:

* Individuals on an unrestricted regular diet with no dietary restrictions (vegan, low FODMAP, gluten free, dairy-free etc) or other fad diets (e.g., keto, intermittent fasting, etc.).
* Healthy subjects will be screened for current or chronic GI symptoms using a 16-item questionnaire.
* Only those with an absence of symptoms will eligible to participate.

Exclusion Criteria:

* For healthy volunteers, will include prior surgery altering the esophagus, stomach, and intestine (except appendectomy).
* Chronic daily use of medications affecting GI secretion or motor function.
* The presence of any GI-motility affecting systemic diseases or untreated psychiatric disease.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Observed Operational Taxonomic Unit (OTU) diversity. | Baseline, Day 56
  Observed OTU counts in each stool sample will be tested at varying cutoffs by determining the number of OTUs per sample.

SECONDARY OUTCOMES:
Adverse Events | 60 days
  Number of participants to report adverse events.
Changes in Shannon diversity index. | Baseline, Day 56
  Observed Shannon diversity index count between PPI and placebo group compare to PPI and probiotic group.
Changes in enrichment according to Kyoto Encyclopedia of Genes and Genomes (KEGG) pathways. | Baseline, Day 56
  Observed changes according to KEGG pathways as compared between PPI and placebo versus PPI and probiotic groups.
Changes in taxa units. | Baseline, Day 56
  Observed changes in taxonomic classifications as compared in PPI and placebo groups versus PPI and probiotic groups.

CONTACTS AND LOCATIONS:
Overall Officials: John DiBaise, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trial Website — https://www.mayo.edu/research/clinical-trials